CLINICAL TRIAL: NCT02462993
Title: EFFECT OF LOCALLY DELIVERED ALOE VERA GEL AS AN ADJUNCT TO SCALING AND ROOT PLANING IN THE TREATMENT OF CHRONIC PERIODONTITIS: A SPLIT-MOUTH CLINICAL AND MICROBIOLOGICAL STUDY
Brief Title: Local Drug Delivery of Aloe Vera Gel in Chronic Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dr. D. Y. Patil Dental College & Hospital (Other)
Responsible Party: Principal Investigator, Santosh Martande, Assistant Professor, Dr. D. Y. Patil Dental College & Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DYPCH/12/PG14
Record Dates: First submitted 2015-05-29; First posted 2015-06-04 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Aloe vera group (Experimental): Group recieving scaling and root planing and aloe vera gel local drug delivery
  Interventions: Drug: Aloe Vera
- SRP group (No Intervention): Group recieving only scaling and root planing

INTERVENTIONS:
Drug: Aloe Vera — Local drug delivery of aloe vera gel
  Arms: Aloe vera group

SUMMARY:
Background: Aloe vera is considered to be the most promising and high-ranking agent as an all-purpose herbal plant amongst herbal agents used in dentistry. This study was designed to evaluate the clinical and microbiological effectiveness of locally delivered aloe vera gel as an adjunct to scaling and root planing in the treatment of chronic periodontitis.

DETAILED DESCRIPTION:
Background: Aloe vera is considered to be the most promising and high-ranking agent as an all-purpose herbal plant amongst herbal agents used in dentistry. This study was designed to evaluate the clinical and microbiological effectiveness of locally delivered aloe vera gel as an adjunct to scaling and root planing in the treatment of chronic periodontitis.

Methods: Twelve subjects diagnosed with chronic generalized periodontitis were selected and randomly divided into two groups: Test group which received scaling and root planning (SRP) followed by application of aloe vera gel as a local drug delivery agent in the deepest periodontal pocket and control group which received SRP alone. Clinical evaluation was undertaken using Plaque index (PI), Gingival index (GI), Probing pocket depth (PPD), Relative attachment level (RAL) and Gingival marginal level (GML) and microbiologic counts (total colony count/ml) were assessed at baseline, 6 weeks and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion in this study was based on the following criteria:

  1. Patients with age group between 30 - 60 years from both sexes.
  2. Chronic periodontitis patients with at least 1 pair of periodontal pocket ≥ 5mm in contra-lateral quadrants.

Exclusion Criteria:

* Exclusion criteria were:

  1. Subjects who have received antibiotic treatment in the preceding 6 months.
  2. Patients with history of prolonged use of antibiotics/ steroids/ immunosuppressive agents /aspirin/ anticoagulants/ other medications including any herbal products.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in Relative Attachment Loss was taken as the primary outcome | 3 months

SECONDARY OUTCOMES:
Change in Probing depth | 3 months
Change in number of microbial species | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Krupa H Pathak, Principal Investigator — Post graduate

REFERENCES:
- [Result] Bhat G, Kudva P, Dodwad V. Aloe vera: Nature's soothing healer to periodontal disease. J Indian Soc Periodontol. 2011 Jul;15(3):205-9. doi: 10.4103/0972-124X.85661. PMID 22028505
- [Result] Perinetti G, Paolantonio M, Cordella C, D'Ercole S, Serra E, Piccolomini R. Clinical and microbiological effects of subgingival administration of two active gels on persistent pockets of chronic periodontitis patients. J Clin Periodontol. 2004 Apr;31(4):273-81. doi: 10.1111/j.1600-051x.2004.00481.x. PMID 15016256